CLINICAL TRIAL: NCT05173207
Title: A Preliminary Investigation of Respiratory-Swallow Coordination in Cardiothoracic Surgical Patients
Brief Title: Respiratory-Swallow Coordination in Cardiothoracic Surgical Patients
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202102635
Record Dates: First submitted 2021-11-12; First posted 2021-12-29 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Thoracic Diseases; Cardiovascular Diseases
Keywords: Dysphagia; Extubation; Respiratory-swallow coordination; Swallow
MeSH Terms: conditions — Thoracic Diseases; Cardiovascular Diseases; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiothoracic surgical patients: Subjects will undergo one simultaneous instrumental examination of swallowing and concurrent monitoring of metrics of respiratory-swallow physiology. Research exam will be performed at bedside within Cardiac & Thoracic Intensive Care Units during their early postoperative recovery.
  Interventions: Diagnostic Test: Videofluoroscopic swallow exam with concurrent monitoring of respiratory-swallow coordination

INTERVENTIONS:
Diagnostic Test: Videofluoroscopic swallow exam with concurrent monitoring of respiratory-swallow coordination — Participants will undergo simultaneous videofluoroscopy, nasal airflow and respiratory inductance plethysmography testing.

SUMMARY:
Dysphagia (swallowing impairment) is a common complication of cardiothoracic surgery (CS). Although alterations in respiratory-swallow coordination is a known underlying pathophysiologic mechanism of dysphagia in multiple patient populations, no group has examined respiratory-swallow physiology in CS patients. The proposed study will examine respiratory-swallow physiology in CS patients and determine its association with unsafe swallowing and inferior health-related outcomes.

DETAILED DESCRIPTION:
The proposed study will examine respiratory-swallow physiology in cardiothoracic surgical patients and determine its association with unsafe swallowing and inferior health-related outcomes. Participation will involve a single postoperative research exam of approximately 60-90 minute duration. Participants will be seated upright and positioned for simultaneous instrumental imaging of swallow physiology, nasal airflow monitoring, and respiratory inductance plethysmography testing.

ELIGIBILITY:
Inclusion criteria:

* Adults over 18 years of age who have undergone cardiothoracic surgery at UF Health
* No allergies to barium
* Not pregnant
* Willing to participate in study

Exclusion criteria:

* Individuals 18 years of age or younger
* Allergies to barium
* Pregnant
* Not willing to participate in study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 individuals undergoing cardiothoracic surgery will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Penetration Aspiration Scale | Up to 1 year
  This scale is a validated measure used by trained blinded clinicians to assign ratings of safety to swallowing bolus trials. The development and use of an 8-point, equal-appearing interval scale (8 being best; 1 being worst) to describe penetration and aspiration events are described. Scores are determined primarily by the depth to which material passes in the airway and by whether or not material entering the airway is expelled.

CONTACTS AND LOCATIONS:
Overall Officials: Emily K Plowman, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No